CLINICAL TRIAL: NCT00828997
Title: Effects of Different Anti-rheumatic Treatments of Arthritis on Antibody Response Following Pneumococcal Vaccination Using Prevenar®
Brief Title: Effects of Different Antirheumatic Treatments of Arthritis on Antibody Response Following Vaccination Using Prevenar®
Acronym: PVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EU-nr 2007-006539-29
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis; Spondylarthropathy
Keywords: rheumatoid arthritis; spondylarthropathy; immunological response following vaccination with Prevenar
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevenar vaccine (Other): all participants are immunized with a dose of pneumococcal conjugate vaccine
  Interventions: Biological: Prevenar vaccination

INTERVENTIONS:
Biological: Prevenar vaccination — vaccination with Prevenar vaccine in patients with arthritis

SUMMARY:
Previous studies have analyzed serological responses following pneumococcal vaccination using 23-valent vaccination (Pneumovax) in Rheumatoid Arthritis (RA) patients that were on different therapeutic modalities including TNF-blockers and methotrexate. The results have shown that serological response was significantly reduced in RA patients receiving methotrexate compared to those receiving TNF-blockers.

In contrast when using polypeptide immunisation (influenza vaccine) we found that anti-TNF significantly impaired the serological response compared to the methotrexate treated RA patients. The aim of this study is to analyze serological responses after Prevenar vaccination in patients with chronic arthritis and to study the impact of different treatment modalities on serological responses.

It will be of interest to see if the result is different compared to the one seen after immunizing with 23-valent nonconjugated pneumococcal polysaccharide vaccine.

DETAILED DESCRIPTION:
Background: Previous studies have analyzed serological responses following pneumococcal vaccination using 23-valent vaccination (Pneumovax) in Rheumatoid Arthritis (RA) patients that were on different therapeutic modalities including TNF-blockers and methotrexate. The results have shown that serological response was significantly reduced in RA patients receiving methotrexate compared to those receiving TNF-blockers (Rheumatology (Oxford) 2006 Jan; 45(1):106-11).

In contrast when using polypeptide immunisation (influenza vaccine) we found that anti-TNF significantly impaired the serological response compared to the methotrexate treated RA patients.

The aim of this study is to analyze serological responses after PREVENAR vaccination in patients with RA or spondylarthropathy and to study the impact of different treatment modalities on serological responses.

It will be of interest to see if the result is different compared to the one seen after immunizing with 23-valent nonconjugated pneumococcal polysaccharide vaccine.

Study design:

Unblinded study in RA patients and patients with spondylarthropathies. All subjects will be vaccinated once with Prevenar and the serological response will be followed by blood draws.

Patient Population to be Included:

RA patients on methotrexate and/or other DMARDS RA patients on anti-TNF drugs as monotherapy RA patients on anti-TNF +MTX and/or other DMARDSs Spondylarthropathy patients on anti-TNF drugs as monotherapy Spondylarthropathy patients on anti-TNF drugs +MTX Spondylarthropathy patients on NSAIDs (There is a possibility to stratify for steroid use).

Primary and Secondary Efficacy Endpoints:

Serological responses to at least 2 pneumococcal serotypes included in Prevenar vaccine between different treatment groups.

An ethical approval from the Ethical Review Board at Lund University is mandatory for this study as well as an approval from the Swedish MPA.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical diagnosis of RA or spondylarthropathy

Exclusion Criteria:

* Pregnancy
* Allergy
* Has received pneumococcal vaccination within 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2008-08; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Serological responses to at least 2 pneumococcal serotypes included in Prevenar vaccine between different treatment groups. | 2009

SECONDARY OUTCOMES:
to analyse if the result is different compared to the one seen after immunizing with 23-valent nonconjugated pneumococcal polysaccharide vaccine. | 2009

CONTACTS AND LOCATIONS:
Overall Officials: Meliha C Kapetanovic, MD,PhD, Principal Investigator — Dept of Rheumatology, Lund University Hospital, Lund, Sweden
Locations (1):
- Lund, Sweden

REFERENCES:
- [Derived] Nagel J, Geborek P, Saxne T, Jonsson G, Englund M, Petersson IF, Nilsson JA, Truedsson L, Kapetanovic MC. The association between antibody levels before and after 7-valent pneumococcal conjugate vaccine immunization and subsequent pneumococcal infection in chronic arthritis patients. Arthritis Res Ther. 2015 May 19;17(1):124. doi: 10.1186/s13075-015-0636-z. PMID 25986458
- [Derived] Nagel J, Geborek P, Saxne T, Jonsson G, Englund M, Petersson IF, Nilsson JA, Kapetanovic MC. The risk of pneumococcal infections after immunization with pneumococcal conjugate vaccine compared to non-vaccinated inflammatory arthritis patients. Scand J Rheumatol. 2015;44(4):271-9. doi: 10.3109/03009742.2014.984754. Epub 2015 Feb 6. PMID 25656734
- [Derived] Crnkic Kapetanovic M, Saxne T, Jonsson G, Truedsson L, Geborek P. Rituximab and abatacept but not tocilizumab impair antibody response to pneumococcal conjugate vaccine in patients with rheumatoid arthritis. Arthritis Res Ther. 2013 Oct 30;15(5):R171. doi: 10.1186/ar4358. PMID 24286269
- [Derived] Crnkic Kapetanovic M, Saxne T, Truedsson L, Geborek P. Persistence of antibody response 1.5 years after vaccination using 7-valent pneumococcal conjugate vaccine in patients with arthritis treated with different antirheumatic drugs. Arthritis Res Ther. 2013 Jan 4;15(1):R1. doi: 10.1186/ar4127. PMID 23286772
- [Derived] Roseman C, Truedsson L, Kapetanovic MC. The effect of smoking and alcohol consumption on markers of systemic inflammation, immunoglobulin levels and immune response following pneumococcal vaccination in patients with arthritis. Arthritis Res Ther. 2012 Jul 23;14(4):R170. doi: 10.1186/ar3923. PMID 22824238
- [Derived] Kapetanovic MC, Roseman C, Jonsson G, Truedsson L, Saxne T, Geborek P. Antibody response is reduced following vaccination with 7-valent conjugate pneumococcal vaccine in adult methotrexate-treated patients with established arthritis, but not those treated with tumor necrosis factor inhibitors. Arthritis Rheum. 2011 Dec;63(12):3723-32. doi: 10.1002/art.30580. PMID 21834061